CLINICAL TRIAL: NCT06639516
Title: Therapeutic Effect of Bifidobacterium Longum in Patients with Acute Pancreatitis: a Randomized, Double-Blind, Placebo-Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Lingyu Luo, Professor, The First Affiliated Hospital of Nanchang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bifidobacterium Longum
Record Dates: First submitted 2024-10-02; First posted 2024-10-15 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Acute Pancreatitis
Keywords: acute pancreatitis; Probiotics
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Bifidobacterium longum capsules (10^10 CFU) twice daily for 14 days
  Interventions: Dietary Supplement: Bifidobacterium longum; Combination Product: Standard clinical treatment
- Placebo group (Placebo Comparator): Placebo capsules twice daily for 14 days
  Interventions: Dietary Supplement: Placebo; Combination Product: Standard clinical treatment

INTERVENTIONS:
Dietary Supplement: Bifidobacterium longum — Bifidobacterium longum
  Arms: Intervention group
Dietary Supplement: Placebo — Placebo
  Arms: Placebo group
Combination Product: Standard clinical treatment — Fasting, gastrointestinal decompression, rehydration, inhibition of pancreatic fluid and pancreatic enzyme secretion, improvement of microcirculation, and support of organ function if organ dysfunction occurs at a later stage (mechanical ventilation, continuous renal replacement therapy, and the use of vasoactive drugs).

SUMMARY:
The purpose of this clinical trial is to investigate the impact of Bifidobacterium longum(BL) on the clinical prognosis of patients with acute pancreatitis(AP), to analyze the correlation between BL and intestinal barrier function, as well as the gut microbiota, and to observe adverse reactions and risks in patients with AP after the use of BL.

Participants will be randomly assigned to two groups: the intervention group and the control group. They will receive:

* Intervention group: Standard clinical treatment + BL capsules (10^10 CFU), twice a day, for a total of 14 days;
* Control group: Standard clinical treatment + placebo capsules, for a total of 14 days.

A total of 60 patients will be included in this study.

DETAILED DESCRIPTION:
Rationale:The impairment of the intestinal mucosal barrier in patients with acute pancreatitis (AP) plays a crucial role in the progression to severe AP(SAP). Our previous research found that the early gut microbiota structure of AP patients is significantly different from that of healthy individuals, characterized by a marked increase in the relative abundance of conditional pathogens such as Escherichia coli and Shigella, while beneficial bacteria that produce short-chain fatty acids, such as Bifidobacterium, are significantly reduced, especially in patients with SAP. Bifidobacterium longum (BL), a well-known probiotic, has been used to treat a variety of diseases. In our previous animal experiments, we found that BL could alleviate pancreatic damage and inflammatory responses in AP mice and regulate the balance of the gut microbiota. Based on these findings, this study aims to assess the impact of BL on the clinical prognosis of AP patients through a randomized controlled trial, in order to provide a scientific basis for the application of BL in the treatment of AP and to further explore its potential clinical value.

Objective: The purpose of this clinical trial is to investigate the impact of BL on the clinical prognosis of patients with AP, to analyze the correlation between BL and intestinal barrier function, as well as the gut microbiota, and to observe adverse reactions and risks in patients with AP after the use of BL.

Study design: Single-center, randomized, double-blind, placebo-controlled study.

Study population:60 adult patients with acute pancreatitis. Intervention: The intervention group receives standard clinical treatment plus BL capsules (10^10 CFU), twice a day, for a total of 14 days; the control group receives standard clinical treatment plus placebo capsules, for a total of 14 days.

Main study parameters/endpoints: The primary endpoint is the number of days without SIRS within 14 days; the secondary endpoints include infectious complications (including fungal infections), parameters related to systemic inflammatory response, intestinal barrier function and gut microbiota composition, indicators related to recovery of intestinal function, antibiotic use, laboratory-related indicators, and clinical outcomes.

Safety: Throughout the study (or afterwards), treatment-emergent adverse events (TEAEs) were recorded, including gastrointestinal adverse reactions (abdominal pain, nausea, vomiting, bloating, or diarrhea) and allergic reactions, and adverse events that led to discontinuation of the study drug were documented.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 year;
2. The diagnosis of acute pancreatitis according to the revised Atlanta classification;
3. The onset time of acute pancreatitis is within 48 hours;
4. APACHE II score of ≥8, or C-reactive protein > 150 mg/L, or SIRS score of ≥3;
5. Signed the informed consent.

Exclusion Criteria:

1. Within 48 hours of onset, there is multi-organ failure;
2. Use of probiotics within the last month;
3. Pancreatitis following endoscopic retrograde cholangiopancreatography (ERCP);
4. Intra-operative diagnosis;
5. Infection/sepsis caused by a second disease;
6. Malignancy;
7. Immunocompromised patients;
8. Pregnancy and/or lactation;
9. Allergy to Bifidobacterium longum.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The number of days without SIRS within 14 days | From randomization to 14 days after treatment
  Patients were randomized into the study group and remained free of SIRS up to 14 days after enrollment, with the total number of SIRS-free days counted

SECONDARY OUTCOMES:
Infectious complications | During the whole study period including follow-up of 90 days
  The occurence of infected pancreatic necrosis, bacteremia, pneumonia, urosepsis, and/or infected ascites，including fungal infections
Intestinal barrier function | Through study completion, an average of 1 year
  Plasma D-lactate(D-lac）
Intestinal barrier function | Through study completion, an average of 1 year
  Diamine oxidase activity(DAO)
Intestinal barrier function | Through study completion, an average of 1 year
  Plasma endotoxin levels
Gut microbiota composition | Baseline , 3 days，7 days and 14 days of treatment
  Fecal samples were collected from patients prior to the start of treatment, as well as on days 3, 7, and 14 after treatment. Subsequently, DNA was extracted from the feces, and the DNA was fragmented by Covaris M220 to screen for fragments of approximately 350 bp to be constructed into paired-end (Paired-End) DNA libraries. Next, libraries were constructed using NEXTFLEX Rapid DNA-Seq. Finally, these libraries were subjected to macro-genomic sequencing for in-depth analysis of microbial community structure and function in the samples.
Systemic inflammatory response parameters (SIRS) | Through study completion, an average of 1 year
  The incidence of persistent SIRS (lasting ≥48 hours)
Systemic inflammatory response parameters (SIRS) | Through study completion, an average of 1 year
  Trends in SIRS score changes
Systemic inflammatory response parameters (SIRS) | Through study completion, an average of 1 year
  Trends in CRP level changes
Gut function recovery-related indicators | Through study completion, an average of 1 year
  Improvement in abdominal signs
Antibiotic usage | Through study completion, an average of 1 year
  The number of days of antibiotic use
Mortality | During the whole study period including follow-up of 90 days
  Occurence of death
(New onset) transient/persistant (multiple) organ failure | During the whole study period including follow-up of 90 days
  The occurence of (new onset) transient/persistant (multiple) organ failure
Disease severity according to the revised Atlanta Classification | During the whole study period including follow-up of 90 days
  Disease severity according to the revised Atlanta Classification
Length of hospital and/or ICU stay | Through study completion, an average of 1 year
  Measured in days
The need (and number of) for surgical, endoscopic or radiologic interventions | During the whole study period including follow-up of 90 days
  The need (and number of) for surgical, endoscopic or radiologic interventions
Readmissions | During the whole study period including follow-up of 90 days
  The occurrence and number of readmissions

CONTACTS AND LOCATIONS:
Overall Officials: Cong He, PhD, Principal Investigator — The First Affiliated Hospital of Nanchang University
Locations (1):
- The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No